CLINICAL TRIAL: NCT00737438
Title: A Phase II Study of Pre-operative Chemotherapy Plus Bevacizumab With Early Salvage Therapy Based on PET Assessment of Response in Patients With Locally Advanced But Resectable Gastric and GEJ Adenocarcinoma
Brief Title: Pre-operative Chemotherapy Plus Bevacizumab With Early Salvage Therapy Based on PET Assessment of Response in Patients With Locally Advanced But Resectable Gastric and GEJ Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-081
Record Dates: First submitted 2008-08-15; First posted 2008-08-19 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: BEVACIZUMAB (AVASTIN); CAPECITABINE (ORAL); CISPLATIN; EPIRUBICIN; IRINOTECAN (CPT-11) CAMPTOSAR; TAXOTERE (DOCETAXEL); ESOPHAGUS; STOMACH; 08-081
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Epirubicin; Cisplatin; Capecitabine; Bevacizumab; Docetaxel; Irinotecan; BaseLine dental cement; Time; Surgical Procedures, Operative

ARMS (1):
- 1 (Experimental): Initial chemo for ALL pts (ECX + BEV): Epirubicin 50 mg/m2 d1 every 21 days Cisplatin 60 mg/m2 d1 every 21 days, Capecitabine 625 mg/m2 po bid days 2-21 (held for 48 hours prior to FDG-PET/CT in week 3) Bev 15 mg/kg d1 every 21 days (cycle 1 & cycle 2 only) Salvage chemotherapy for metabolic non-responders (DI + BEV): Docetaxel 30 mg/m2 d1, d8 every 21 days, CPT-11 50 mg/m2 d1, d8 every 21 days, Bev 15 mg/kg d1, cycle 2 only 2 cycles are planned prior to resection.
  Pts who aren't Cisplatin candidates (i.e. Creatinine clearance 40-60/cc, older age, marginal PS,etc.) may get oxaliplatin instead of cisplatin after discus with the PI. Oxaliplatin will be admin at 130 mg/m2 on day 1 every 21 days. Pts who aren't able to get Capecitabine (i.e. insurance restriction, unable to swallow, etc.) may get infusional fluorouracil instead of capecitabine after discus with the PI. Fluorouracil will be admin at 200 mg/m2/d x 21 days (held for 48 hours prior to FDGPET/ CT scan in week 3 of cycle 1).
  Interventions: Drug: epirubicin, cisplatin, capecitabine, bevacizumab, docetaxel and irinotecan

INTERVENTIONS:
Drug: epirubicin, cisplatin, capecitabine, bevacizumab, docetaxel and irinotecan — Patients with FDG avid locally advanced but resectable gastric or GEJ adenocarcinoma will receive preoperative therapy with epirubicin, cisplatin, capecitabine (ECX), and bevacizumab. Each cycle of therapy is 21 days. Near the completion of cycle 1 of therapy (eg during week 3, target days 18-21), patients will undergo a second FDG-PET/CT scan. Note, patients will hold capecitabine for 48 hours prior to the FDG-PET/CT scan.
  Patients with a good metabolic response (eg. > 35% reduction in FDG uptake at the primary tumor on the week 3 PET scan as compared with baseline FDG uptake) will continue ECX for 2 additional cycles (cycle 2 and 3).
  Cycle 2 will be administered with bevacizumab and cycle 3 will be administered without bevacizumab. Patients will then proceed to surgery approximately 4-6 weeks following the completion of cycle 3. There is a 10-12 week time interval (eg. 70-84 days) between the last bevacizumab treatment and surgery.
  Other Names: Patients who have a poor PET response to cycle 1 of ECX plus bevacizumab; (eg. < 35% FDG reduction on the week 3 PET scan compared with baseline); will be switched to salvage therapy of docetaxel and irinotecan (DI).; This treatment will be administered on week 1 and 2 of a 3; week cycle for 2 cycles. Patients will receive bevacizumab for the 1st cycle; of salvage docetaxel/irinotecan only. There is again a planned 10-12 week time; interval (eg. 70-84 days) between the last bevacizumab treatment and surgery.

SUMMARY:
This study is being done to find out how effective a new treatment strategy is on your cancer. In this strategy, the response your tumor has to the first cycle of therapy will help select the next treatments. We also will find out the effects, both good and/or bad, a drug called bevacizumab has on you and your tumor when given with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have microscopically confirmed adenocarcinoma of the stomach or GE junction. Tumors involving the GE junction must have the bulk of their disease in the stomach; tumors of the distal esophagus that extend less than 2cm into the stomach are ineligible for this study.
* All patients must be considered candidates for surgical resection.
* Patients must have FDG-avid malignancies.
* FDG avid tumors are defined as primary tumors with an increased tracer uptake in the region of the tumor that has an SUV > or = to 3.5 or a tumor:liver ratio > or = to 1.5, and felt to be "probably" or "definitely malignant" (i.e. likelihood score of 3 or 4) by the reference nuclear medicine physician.
* All patients must have localized cancer potentially curable by surgery. The tumor stage should be T any N+ M0 or T3-T4a N any M0(AJCC 7th Edition), by staging that includes a CT scan and either laparoscopy or endoscopic ultrasound. Patients with T1-2 N0M0 or patients with distant metastatic disease (i.e. M1) are ineligible. Any sites of suspected M1 disease by these criteria must be proven to be M0 prior to entrance into the neoadjuvant study.
* Patients may not have received prior chemotherapy or radiation for this disease.
* The patient is at least 18 years of age.
* If female and of child bearing potential, the patient has a negative serum pregnancy test within 14 days of starting therapy, and, if male or female and of child bearing potential, currently uses (and agree to continue to use throughout the study) an acceptable method of birth control (IUD, oral contraceptive, or barrier device). They should agree to continue to use these for three months after the study is completed. The patient also agrees to refrain from nursing during the duration of the study and for at least two months after the study is completed. Pregnant or lactating females are not included because the anti-proliferative effects of bevacizumab may be harmful to the fetus or developing infant.

Karnofsky performance status > or = to 70%.

* The patient has adequate hematopoietic function, defined as having a total neutrophil count (ANC) ≥ or = to 1500/mm3, a platelet count ≥ or = 100,000/mm3. The patient has adequate renal and hepatic function, defined as having a serum creatinine ≤ or = to 2.5 mg/dl, urinalysis demonstrating < 2+ proteinuria and/or a urine protein/creatinine (UPC) ratio < 1.0. LFTs include a total serum bilirubin ≤ than or = to 2 x ULN, serum AST (SGOT)/ALT (SGPT) and ALK PHOS < than or = to 2.5 ULN.
* The patient has a PT (INR) < than or = to 1.5 and an PTT < than or = to 3 seconds above the upper limits of normal (i.e. at MSKCC PTT < than or = to 37.7 sec) if the patient is not on anticoagulation.
* If a patient is on full-dose anticoagulants, the following criteria should be met for enrollment

  1. If using warfarin, the subject must have an in-range INR (usually between 2 and 3) and on a stable dose of warfarin.
  2. The subject must not have active bleeding or pathological conditions that carry high risk of bleeding (e.g. tumor involving major vessels, known varices).
* Ability to understand informed consent and signing of written informed consent document prior to the initiation of treatment.

Exclusion Criteria:

* Any metastatic disease.
* Significant cardiac disease as defined as:
* New York Heart Association (NYHA) grade II or greater (see Appendix B for NYHA Class),
* congestive heart failure, or history of myocardial infarction or unstable angina within 12 months of study enrollment
* Any history of stroke or transient ischemic attack at any time.
* Pregnant (positive pregnancy test) or lactating women. A pregnancy test will be performed on sexually active women of childbearing potential prior to entry into the study. Treatment may not begin until the results of the pregnancy test are ascertained.
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) on antihypertensive therapy.
* Any prior history of hypertensive crisis or hypertensive encephalopathy.
* Significant vascular disease (e.g. aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease (ie. grade 2 or higher).
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting therapy (eg. day 0).
* Core biopsy or other minor surgical procedure, excluding placement of a vascular device, within 7 days of starting therapy.
* Evidence of bleeding diathesis or coagulopathy.
* Proteinuria at screening as demonstrated by either

  * Urine protein:creatinine (UPC) ratio > 1.0 at screening, or
  * Urine dipstick for proteinuria > or = to 2+ (patients discovered to have > or = to 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hour urine collection and must demonstrate < than or = to 1g of protein in 24 hours to be eligible).
* Serious intercurrent infections, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment.
* Serious, non-healing wound, ulcer, or bone fracture.
* Grade 2 or greater pre-existing peripheral neuropathy.
* Psychiatric disorders rendering patients incapable of complying with the requirements of the protocol.
* Any concurrent active malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer or carcinoma-in-situ of the uterine cervix. Patients with previous malignancies but without evidence of disease for > 5 years will be allowed to enter the trial.
* Clinically significant hearing loss.
* EKG evidence of acute ischemia or significant conduction abnormality, as determined by the treating physician.
* Known hypersensitivity to Chinese hamster ovary cell products, other recominant human antibodies, or to any component of bevacizumab.
* Patients with any other medical condition or reason that, in the investigator's opinion, makes the patient unsuitable to participate in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ilson, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center, Commack, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: ALL patients - Pre-operative Chemotherapy Plus Bevacizumab with Early Salvage Therapy in Patients with Locally Advanced but Resectable Gastric and GEJ Adenocarcinoma
Period: Overall Study
Arm/Group | All Patients
Started | 23
Completed | 20
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Patient ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Will be Characterized by the Patient's FDG-PET Scan
Description: A good early FDG Response is a reduction in FDG uptake on the week 3 PET scan of > or = to 35% from baseline. An FDG PET non-responder will be defined as having a decrease of < 35% on the week 3 PET scan compared with baseline.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 20
participants
  Metabolic Responder | 11
  Non-Metabolic Responder | 9

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 12/23
Other Adverse Events (participants affected / at risk) | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=23)
Anorexia (General disorders) | 1 (1)
Death not associated with CTCAE term- Death NOS (General disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Fistula, GI- Stomach (Gastrointestinal disorders) | 1 (1)
Infection with Grade 3/4 neutropenia, Lung (pneumonia) (Infections and infestations) | 1 (1)
Leak, GI- Small Bowel (Gastrointestinal disorders) | 1 (1)
Leak, GI- Stomach (Gastrointestinal disorders) | 1 (1)
Mucositis (Clincal exam)- Oral cavity (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 1 (1)
Pain - Abdomen NOS (General disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Thrombosis/embolism (vascular access-related) (Cardiac disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight loss (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=23)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 11
Alkaline phosphatase (Metabolism and nutrition disorders) | 2
ALT, SGPT (Blood and lymphatic system disorders) | 4
Anorexia (General disorders) | 7
AST, SGOT (Blood and lymphatic system disorders) | 4
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 5
Creatinine (Metabolism and nutrition disorders) | 4
Dehydration (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 7
Fatigue (asthenia, lethargy, malaise) (General disorders) | 13
Fever (in the absence of neutropenia) (General disorders) | 3
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 12
Glucose, low (hypoglycemia) (Metabolism and nutrition disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 16
prothrombin time international normalized ratio (Blood and lymphatic system disorders) | 2
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 12
Lymphopenia (Blood and lymphatic system disorders) | 8
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 3
Mucositis - Larynx (General disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 14
Pain - Abdomen NOS (General disorders) | 5
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 10
Platelets (Blood and lymphatic system disorders) | 2
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 2
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 5
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2
Sodium, high (hypernatremia) (Metabolism and nutrition disorders) | 2
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 3
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes